# Longitudinal Study of Dental Implant Therapy in HIV Positive Patients

Study Protocol & Statistical Analysis Plan

NCT01211288

August 30, 2019

Toni Tien Neumeier, DMD, Principal Investigator University of Alabama at Birmingham Birmingham, AL 35294



#### APPENDIX 1

Protocol

D-2007-51

## PROTOCOL SYNOPSIS

#### Title

Longitudinal Study of Dental Implant Therapy in HIV Positive Patients

Investigator (Insert here the name, mailing address, email address, and phone number of the Coordinating Investigator (for multi-centre studies) or the Principal Investigator (for single-centre studies))

A. Principle Investigator:

Toni Tien Neumeier, MS, DMD, FAGD, FACD

Prosthodontist, Associate Professor, UAB Comprehensive Dentistry Department

1919 7th Ave South, SDB 530

Birmingham, AL 35294

Neumeier@uab.edu

205-934-5459

- B. Co- Investigators:
  - 1. Jeff Hill, DMD

General Dentist, Assistant professor, Director 1917 HIV/AIDS Dental Clinic, UAB Comprehensive Dentistry Department

2. Mike Edwards, DMD, FAGD, MAGD

Assistant clinic professor, UAB Comprehensive Dentistry Department Private Practice General Dentistry, Wedowee AL.

3. Perng - Ru Liu, DDS, MS, DMD

Prosthodontist, Professor and Chair, UAB Comprehensive Dentistry Department

4. Lance Ramp, DMD, PHD

Prosthodontist, Associate Professor, UAB Comprehensive Dentistry Department

5. Richard Weems, DMD

Radiologist, Associate Professor, Director of Clinical Operations and Dental Radiology, UAB Diagnostic Science Department

6. Patricia Devilliers, DDS, MS

Oral and Maxillofacial Pathologist, Assistant Professor, UAB Anatomic Pathology Department

<<>>

Study centre(s) and number of subjects planned (Insert here the address where the study will be conducted, number of patients planned and if applicable distribution of patients per site)

UAB School of Dentistry
Department of Comprehensive Dentistry
1919 7<sup>th</sup> Ave South
Birmingham, AL 35294





Total 40 patients will be treated in the 2<sup>nd</sup> floor main clinic

20 HIV (+) patients will be selected from the 1917 Dental Clinic and 20 patients will be selected from UAB School of Dentistry patients.

2. Cone Beam CT scanned at UAB School of Dentistry Periodontal research clinic

<<>>

Study period

<<Month and year>>

<<Month and year>>

Estimated Start date and End date

January 2010

December 2014

Date of first data available for presentation

December 2011

Objectives (Insert objectives)

- 1. To study the short term and long term osseous integration of implant supported restorations on immunocompromised (HIV positive) patients.
- 2. Radiographic examination of implant osseous integration using Cone Beam CT and traditional vertical bitewing radiographs.
- 3. Histologic examination of bone biopsies from each implant surgical site, at the time of initial placement, and from failing implant sites, including histologic examination of the implant-bone interface.

Study design (Insert a one-sentence summary of study design features

Provide HIV (+) patients with implant supported restorations, using HIV (-) patients as controls.

<<>>

Target patient population (Insert a description of target population and indication studied)

20 HTV (+) patients with the following requirements:

Age 19 and older,

Hemoglobin >8g/dl, Absolute neutrophil count >750/mm3, Platelet count>75,000cells/mm3, AST< 5 times the upper limit of normal (ULN),

Bilirubin < 2.5 times ULN, Alkaline phosphate < 5 times ULN, Creatinine < 2.5 mg/ml

Non-smoker (quite smoking at least 6 months)

Controlled Type II diabetes

Controlled hypertension

Non bisphosphate user

Non-bruxer

Misch Available Bone classification divisions A, B, C

Misch Bone Density classification D1, D2, D3

Minimal available bone width 5mm

Minimal available bone height 10mm

Minimum bone graft with freeze dried demineralised bone upon implant placement

Extraction site has to be healed up for minimum 3 months for mandibular and 6 months for maxillary before implant placement

Flap or flapless implant placement with surgical stent as guidance

Implant supported restorations are limited to the following edentulous areas:

Mandibular arches, excluding 3<sup>rd</sup> molar areas

Maxillary anterior and premolar areas

Exclude extensive bone graft involvement and sinus lift

No immediate implant loading

The



Total numbers of implant restorations are limited to;

Maximum of 4 units of fixed prosthesis with minimum 2 implants support for maxillary and mandibular anterior region,

3 units bridge with 2 implant supports,

2 units bridge with 2 implant supports,

Single implant support crown

Permanent implant restoration 3 months after implant placement for mandibular and 6 months for maxillary.

All implant supported restorations will be cement-retained restorations.

Dental material: either full metal restoration or porcelain fused with metal restoration.

20 HIV-negative patients following the same requirements as above.

Investigational product/comparator (State the devices / products that will be investigated / / used and for comparative studies also the comparator/s)

- 1. Cone beam CT full facial scan on every patient before and after implant placement on surgical site single arch at 1 year, 2 year, 3 year follow up (i-CAT \$600 per patient x40 =\$ 24,000)
- 2. Facilitate Pro software convert Dicom images for implant placement design and surgical stent fabrication (\$12,000)
- 3. Surgical tools for implant placement:

(syringe, needles, elevators, periotomes, extraction forceps #150 & #151, bone spreading chisels, bone grinder, bone trap, bone compactor, bone curette, osteotomes, resorbable and non-resorbable sutures, needle holders, scissors

Surgical stent, two surgical bundles, two surgical trays, one surgical motor, two surgical handpiece heads, two full restorative trays and bundles, surgical saline bags for surgical

irrigation, disposable irrigation kits for drill unit, disposable drills. Pulse oximetry) (\$ 30,000)

- 4. Root form implants of various sizes, cover screws (\$250 per implant x est. 80=\$20,000)
- 5. Freeze dried demineralised bone as bone graft material (\$ 100/ 0.5cc vial x est.20 = \$ 2,000) (\$ 100/ membrane x est. 20 = \$ 2,000)
- 7. Poly vinyl siloxane impression materials (\$4,000)
- 8. Prosthodontic instrument kits plus laboratory fee (impression transfer material, implant abutments, implant analogues, Cresco Precision system)

(\$ 400 per implant restoration x est. 80 = \$32,000)

9. Two WhipMix Semi- adjustable articulators

 $(\$ 800 \times 2 = \$1,600)$ 

10. Half-time patient coordinator

(\$ 18,000 or neg.)

\*11. Computer for information storage and portable printer

(\$ 3,000)

12. SLR camera with Macro-lens and flash

- (\$2,500)
- Histological examination of 40 bone biopsies processed at UAB Anatomic Pathology Lab,
   including special stains and decalcification (\$ 8,000
- 14. Processing of failed implants at the UAB Bone Core facility with subsequent histologic examination of implant-bone interface (\$200.00 per failed implant x est. 5 =\$1,000)
- 15. Journal publication expenses

(\$2000.00)

16. Travel expenses to national and/or international meetings by the PI investigator and one co-investigator (\$ 4000.00)

Total budget: \$166,000

iFC



Outcome variables (Indicate which variable is the primary variable for the study)

Efficacy (List all efficacy variables and indicate clearly your primary outcome variable

The primary variable examined will be the treatment outcome as measured according to the Albrektsson and Zarb criteria for implant success. Patients will be examined at each interval for the presence of pain, infection, mobility, and radiographic bone height of each implant

Additional clinical assessments (Describe use of any additional clinical assessments e.g. clinical photographs etc.

- 1. All selected patients will have prior medical authorization to have surgical procedure performed. Patients with undergo complete oral clinical examination as well as cone beam CT scan, selected periapical and vertical bitewing radiographs on planning implant placement site, full mouth photography, diagnostic casts, and surgical stint before implant placement.
- 2. Cone Beam CT on the implant sites of arches at 1 year, 2 years and 3 years post placement follow-up (Cone Beam CT provides 1:1 ratio image, view in 3- dimensions, limited radiation exposure). The images will be evaluated by the dental radiologist.

Compare accuracy and efficiency of Cone Beam CT image of alveolar bone around implant in 3dimensions vs. of conventional standard X-ray examination of bone lost around implant in 2dimensions.

- 3. Histologic examination of the bone biopsy from the implant sites will provide scientific evidence of the bone changes that may occur in the process of implant osteointegration under immunocompromised conditions.
- 4. Photograph during implant restoration procedure and after complete restoration.
- 5. Patient post-implant restoration survey (such as: general satisfaction, social life, mastication on hard food, comfort).

Statistical methods (Describe as relevant the statistical methods to be used, the populations to be analysed (e.g. intention to treat, per-protocol), and any interim analyses)

Descriptive statistics will be applied to acquire the mean parameter values, range, and implant success rate as determined by the Albrektsson and Zarb criteria.

With rigorous inclusion/exclusion criteria proposed, parametric data will be analysed using ANOVA methods. Nonparametric (yes/no) criteria will be analyzed with the Chi-Square method.

Publications / Presentations (Describe your plans with regard to publications or public presentations i.e. what journals or conferences/meetings)

Peer reviewed journals such as: Journal of American Dental Association, Journal of Prosthodontics, Journal of General Dentistry.

Oral platform presentations at various national and international dental meetings at Astra's discretion

BL-MC-0804-B

D-2007-051FINAL20091217

12(16)



## APPENDIX 2 - Details of products to be provided:

Investigator name: Toni Neumeier, UAB

Study Title: Longitudinal Study of Dental Implant Therapy in HIV Positive Patients

Astra Tech reference no.: D-2007-51

| Product | Ref. no. | Quantity |
|---------------------------------|----------|----------|
| Restorative Instrument Kit | 24879 | 2 |
| Restorative Tray | 22495 | 2 |
| Torque Wrench Kit | 24100 | 2 |
| Torque Wrench Bit, Locator-15mm | 24490 | 2 |
| Wrench Adapter | 24572 | 2 |
| Implant Unit SI-915, 115 V | 24360 | 2 |
| Cont Ang.W&H WS-75 E/KM AE | 22903 | 2 |
| Surgical Instrument Kit | 24878 | . 2 |
| Driver Handle | 24358 | 2 |
| Surgical Tray | 24349 | 2 |
| Ratchet Wrench | 24357 | 2 |
| Hex Screwdriver, Short | 22514 | 4 |
| Hex Screwdriver, Intermediate | 22515 | 4 |
| Osteotome Kit | 22956 | 2 |
| SP Drill Kit, Short | 22898 | 24 |
| SP Drill Kit, Long | 22899 | 24 |
| SP Twist Drill, 3.35 mm, Short | 22908 | 12 |
| SP Twist Drill, 3.35 mm, Long | 22909 | 12 |
| SP Twist Drill, 3.7 mm, Short | 22910 | 24 |
| SP Twist Drill, 3.7 mm, Long | 22911 | 24 |
| SP Conical Drill, 4.5mm, Short | 22921 | 24 |
| SP Conical Drill, 4.5mm, Long | 22922 | 24 |
| SP Conical Drill, 5.0mm, Short | 22923 | 24 |
| SP Conical Drill, 5.0mm, Long | 22924 | 24 |
| OsseoSpeed 3.5 S - 9 mm | 24611 | 8 |
| OsseoSpeed 3.5 S - 11 mm | 24612 | 8 |
| OsseoSpeed 3.5 S - 13 mm | 24613 | 8 |
| OsseoSpeed 4.0 S - 9 mm | 24621 | 8 |
| OsseoSpeed 4.0 S - 11 mm | 24622 | 10 |
| OsseoSpeed 4.0 S - 13 mm | 24623 | 8 |
| OsseoSpeed 4.5 - 9 mm | 24631 | 8 |
| OsseoSpeed 4.5 - 11 mm | 24632 | 10 |
| OsseoSpeed 4.5 - 13 mm | 24633 | 8 |
| OsseoSpeed 5.0 - 9 mm | 24641 | 8 |





| OsseoSpeed 5.0 - 11 mm | 24642 | 8 |
|---------------------------------|-------|-----|
| OsseoSpeed 5.0 - 13 mm | 24643 | 8 |
| Implant Transfer 3.5/4,0 Short | 24547 | 30 |
| Implant Transfer 3.5/4.0 Long | 24548 | 20 |
| Fixt. Transfer 4.5/5.0,Short | 22433 | 30 |
| Fixt. Transfer 4.5/5.0, Long | 22485 | 20 |
| Implant Replica 3.5/4.0 | 24276 | 50 |
| Implant Replica 4.5/5.0 | 22509 | 50 |
| Ti-Zir Design 3.5/4.0 Try-in | 24847 | 4 |
| Ti-Zir Design 4.5/5.0 Try-in | 24849 | 4 |
| TiDesign 3.5/4.0 - @ 5.5, 1.5mm | 24287 | 12 |
| TiDesign 3.5/4.0 - Ø 5.5, 3mm | 24288 | 12 |
| TiDesign 4.5/5.0 - 05.5,1.5 mm | 24235 | 12 |
| TiDesign 4.5/5,0 -05.5, 3mm | 24236 | 12 |
| ZirDesign 3.5/4.0 @ 4.5 1.5 mm | 24702 | 8 |
| ZirDesign 3.5/4.0 Ø 5.5 1.5 mm | 24704 | 8 |
| ZirDesign 4.5/5.0 Ø 5.5 1.5 mm | 24707 | 8 |
| ZirDesign 4.5/5.0 @ 5.5 3 mm | 24708 | В |
| Dir.Abutm.API 3.5/4.0-Ø5, 1mm | 24555 | 4 |
| Dir.Abutm.API 3.5/4.0-@5.2.5mm | 24556 | 4 |
| Dir.Abutm.API 4.5/5.0-Ø5, 1mm | 24559 | 4 |
| Dir.Abutm.API 4.5/5.0-@5,2.5mm | 24560 | 4 |
| Dir.Abutm.API 4.5/5.0-@6, 1mm | 24562 | 4 |
| Dir.Abutm.API 4.5/5.0-@6,2.5mm | 24563 | 4 |
| Cover Screw 3.5/4.0 - 0 mm | 24328 | 40 |
| Cover Screw 4.5/5.0 - 0mm | 24447 | 40 |
| Healing Abutm.3.5/4.0-@4,2mm | 24574 | 12 |
| Healing Abutm.3.5/4.0-04.5,4mm | 24575 | 12 |
| Healing Abutm.3.5/4.0-@5.5,2mm | 24577 | 12 |
| Healing Abutm.3.5/4.0-05.5,4mm | 24578 | 12 |
| Healing Abutm.4.5/5.0-@5.5,2mm | 24582 | 12 |
| Healing Abutm.4.5/5.0-@5.5,4mm | 24583 | 12 |
| Healing Abutm.4.5/5.0-@6.5,2mm | 24585 | 12 |
| Healing Abutm.4.5/5,0-@6.5,4mm | 24586 | 12 |
| Bone Trap | 22179 | 8 |
| Disposable Irrigation Set | 22176 | . 8 |
| Periotome,straight/curved edge | 24274 | 2 |
| Periotome, curved/straight | 24275 | 2 |
| Grinding Handle | 22740 | 2 |
| Bowl, Titanium | 22137 | 4 |
| Forceps 94 | 22437 | 4 |

BL-MC-0804-8



| Facilitate Instrument Kit | 24819 | 2 |
|--------------------------------|-------|---|
| Direct Abutment 3.5/4.0 Try-in | 24848 | 4 |
| Direct Abutment 4.5/5.0 Try-in | 24850 | 4 |

Products will be distributed to the below contact person and address: Dr. Toni Tien Neumeier Comprehensive Dentistry Department 1919 7th Ave South SDB 530 Birmingham, Al 35294

